CLINICAL TRIAL: NCT04406337
Title: A Comparative Study of Low Intensity Pulsed Ultrasound (Osteotron IV) Versus High Intensity Continuous Ultrasound Therapy in Knee Osteoarthritis
Brief Title: Low Intensity Pulsed Ultrasound Versus High Intensity Continuous Ultrasound Therapy in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health and Sports, Myanmar (Other Government)
Collaborators: University of Medicine 1 Yangon (Other); Physical Medicine and Rehabilitation, Yangon General Hospital (Unknown)
Responsible Party: Principal Investigator, Wunn Lei Thwe, Principal Investigator, Ministry of Health and Sports, Myanmar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMR
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis; Rheumatic Diseases; Musculoskeletal Diseases
Keywords: Low intensity pulsed ultrasound (LIPUS); High intensity continuous ultrasound; Knee pain; Knee stiffness; Randomized controlled trial; Myanmar; Osteotron
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Rheumatic Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity pulsed ultrasound (Experimental): Participants in this arm will receive low intensity pulsed ultrasound therapy on the affected knees for 20 minutes per day, 5 days a week for 4 weeks. Conventional physiotherapy of quadriceps muscle exercise and health education about life style will also be given.
  Interventions: Device: Low intensity pulsed ultrasound
- High intensity continuous ultrasound (Active Comparator): Participants in this arm will receive high intensity continuous ultrasound therapy on the affected knees for 10 minutes per day, 5 days a week for 4 weeks. Conventional physiotherapy of quadriceps muscle exercise and health education about life style will also be given.
  Interventions: Device: High intensity continuous ultrasound

INTERVENTIONS:
Device: Low intensity pulsed ultrasound — Low intensity pulsed ultrasound therapy will use ultrasound with frequency of 1.5 MHz, power intensity of 30 mW/cm^2 (0.03 W/cm^2 ) and 20% duty cycle.
  Other Names: Osteotron IV
  Arms: Low intensity pulsed ultrasound
Device: High intensity continuous ultrasound — High intensity continuous ultrasound therapy will use ultrasound with frequency of 1 MHz, power intensity of 3 W/cm^2 and 100% duty cycle.
  Other Names: US 50 (Medical Italia)
  Arms: High intensity continuous ultrasound

SUMMARY:
To compare the effects of low intensity pulsed ultrasound with high intensity continuous ultrasound in knee osteoarthritis

DETAILED DESCRIPTION:
Knee osteoarthritis is a common disorder affecting elderly and obese. Currently, there are 3 types of treatment; pharmacological, non-pharmacological and surgery. Though ultrasound, a non-pharmacological treatment, is increasingly used in knee osteoarthritis, the advantages and disadvantages of low intensity pulsed ultrasound (LIPUS) and high intensity continuous ultrasound (HICUS) are yet to be clarified. Therefore, a randomized control trial will be done to compare LIPUS and HICUS in participants with knee osteoarthritis presenting to Department of Physical Medicine and Rehabilitation, Yangon General Hospital, Myanmar.

ELIGIBILITY:
Inclusion Criteria:

* Participants with knee pain (VAS 3 to 6)
* Kellgren and Lawrence grade 2 and 3 in X' ray knee joint

Exclusion Criteria:

* Rheumatoid arthritis, Gouty arthritis, Spondyloarthropathies, Metabolic arthropathies
* Infection of knee joint
* Tumor of knee joint
* History of hypersensitivity to heat
* Previous knee surgery in affected side
* Intra-articular injection within previous 3 months
* Participants taking treatment with other physical modalities such as low-level laser therapy and Trans Cutaneous Electrical Nerve Stimulation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 8 weeks
  It is one of the most commonly used measures of pain intensity and it is divided into 10 ordinal ratings with 0 being "no pain" and 10 being "pain as bad as it could be".
Western Ontario McMaster University Osteoarthritis Index Inventory (WOMAC) | 8 weeks
  This index measures clinically important symptoms of pain, stiffness and function. It consists of 23 questions (5 pain, 2 stiffness and 16 physical function) and the maximum score is 100, indicating the worst outcome while the minimum score is 0, indicating the best outcome.
Percentage of participants with skin irritation | 8 weeks
  Skin irritation, a possible complication of ultrasound therapy, will be recorded as a dichotomous variable (i.e. present or absent).
Percentage of participants with tingling | 8 weeks
  Tingling sensation, a possible complication of ultrasound therapy, will be recorded as a dichotomous variable (i.e. present or absent).
Percentage of participants with oedema | 8 weeks
  Oedema, a possible complication of ultrasound therapy, will be recorded as a dichotomous variable (i.e. present or absent).
Percentage of participants with burns | 8 weeks
  Burns, a possible complication of ultrasound therapy, will be recorded as a dichotomous variable (i.e. present or absent).

CONTACTS AND LOCATIONS:
Overall Officials: Khin Myo Hla, PhD M.B.,B.S, Study Chair — Physical Medicine and Rehabilitation Department, Yangon General Hospital; Soe Soe Khaing, PhD M.B.,B.S, Study Director — Physical Medicine and Rehabilitation Department, Yangon General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Yangon General Hospital, Yangon, Burma

IPD SHARING:
Plan to Share IPD: No